CLINICAL TRIAL: NCT02088827
Title: Effects of Sedentary Behaviour on Metabolic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kenneth Madden, Head, VGH Division of Geriatric Medicine, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H13-01886
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Sedentary Lifestyle; Type 2 Diabetes
Keywords: Exercise; Sedentary Behaviour; Type 2 Diabetes; Older Adults
MeSH Terms: conditions — Sedentary Behavior; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activity (Other): During a 4 hour Meal Test subjects will cycle for 2 minutes every 20 minutes
  Interventions: Other: Activity
- Inactivity (Other): During a 4 hour Meal Test study subjects will remain inactive (remain lying on a bed)
  Interventions: Other: Inactivity

INTERVENTIONS:
Other: Inactivity — Subjects will remain inactive (lying on a bed) for 4 hours.
  Arms: Inactivity
Other: Activity — Subjects will spend 4 hours of inactivity (lying on a bed) broken up by 2 minutes of moderate intensity biking (on a stationary bike) every 20 minutes.
  Arms: Activity

SUMMARY:
The rates of sedentary activity are increasing. Studies have shown that time spent on doing sedentary activities is an independent risk factor for cardiovascular disease. Prior studies have shown that interrupting inactivity improved the body's handling of blood glucose and gene expression. The investigators plan to explore this further by examining the effects of interrupting 4 hours of inactivity with 2 minutes of moderate intensity exercise every 20 minutes on the following metabolic parameters: blood pressure, cortisol, C-Reactive Protein, glucose and insulin levels.

DETAILED DESCRIPTION:
There is a current trend towards increasing time spent in sedentary behaviour. More jobs are being automated, and more time is spent in front of a computer, playing video games and watching television.Current studies suggest that sedentary behaviour is an independent risk factor for cardiovascular disease. Increasing time spent in sedentary behaviour has been linked to all-cause mortality, markers of cardiovascular disease and metabolic syndrome. However, the data is mainly from cross-sectional studies and based on self-recall, limiting the ability to draw definitive conclusions.

Current exercise guidelines recommend at least 150 minutes of moderate to vigorous intensity exercise per week. It may be difficult for some elderly people to meet these guidelines. Older adults with diabetes are already at a higher risk fo conditions that are affected by sedentary behaviour and may stand to benefit the most from intervention.

This study proposes to study the effects of breaking up sedentary activity with moderate intensity exercise on multiple metabolic parameters in older adults with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* type 2 diabetes managed with diet or oral hypoglycemic agents

Exclusion Criteria:

* using insulin to manage diabetes
* baseline of pre-session blood glucose reading equal to or greater than 10 mmol/L
* any medical condition that would limit the ability to perform activity portion of the study
* people not comfortable exercising on a stationary bicycle
* subject answers yes to one of more of the questions in the Physical Activity Readiness Questionnaire

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | every 60 minutes for 4 hours

SECONDARY OUTCOMES:
C Reactive Protein | every 60 minutes for 4 hours
Insulin Levels | every 60 minutes for 4 hours
Blood glucose levels | every 60 minutes for 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Madden, MSc, MD, Principal Investigator — University of British Columbia
Locations (1):
- Gerontology Research Lab, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No